CLINICAL TRIAL: NCT06390449
Title: Investigation of the Effect of the Use of Web 2.0 Tools in Nursing Education on the Development of Student Web Pedagogical Content Knowledge: Randomized Controlled Trial
Brief Title: The Impact of Web 2.0 Tools on Nursing Education
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erzurum Technical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: NM:11.23.ND:19.10.2023
Record Dates: First submitted 2024-03-22; First posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Educational Problems

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): "Kahoot application", which is in the digital test category as a Web 2.0 tool, will be applied after teaching the basic principles and practices in nursing course for 6 weeks. After the applications are completed, the personal information form and the "Web Pedagogical Content Knowledge Scale" will be applied again to both groups.
  Interventions: Other: Kahoot intervention
- Control (No Intervention): The students in the control group will be taught only basic principles and practices in nursing for 6 weeks. The study will be carried out without using the WEB 2.0 tool. After the applications are completed, the personal information form and the "Web Pedagogical Content Knowledge Scale" will be applied again to both groups.

INTERVENTIONS:
Other: Kahoot intervention — Kahoot, one of the WEB-2.0 tools, will be applied to students who are second-year students of the nursing department and taking the basic principles and practices in nursing course after the course.
  Arms: Experimental

SUMMARY:
This research was planned experimentally to investigate the effect of teaching supported by WEB 2.0 tools on the development of WEB pedagogical content knowledge of nursing students. Innovative learning technologies provide easy and fast access to information. One of the important opportunities provided by the Internet is that it facilitates the transfer of information in education and enables active learning thanks to WEB 2.0 applications.

The use of WEB 2.0 tools in nursing education provides significant benefits to the cognitive, affective and behavioral fields. Considering their important role in education, academic nurses' technological applications are critical to achieve good results in this context. For this reason, it is very important to shed light on the use of Web 2.0 tools for nursing education, to enlighten nurse candidates about the general use of Web 2.0 tools, and at the same time to discover the best technological practices they use.

DETAILED DESCRIPTION:
In this study, a priori power analysis was performed before starting the study to determine the sample size. In the power analysis, it was determined that the number of samples should be 80, 40 interventional and 40 control, with a 0.05 significance level, 95% confidence interval, 95% power and a 5% margin of error.

SPSS 23.0 (Statistical Program for Social Sciences) package program will be used to evaluate the data obtained from the research. The suitability of variables to normal distribution will be examined visually (histograms, probability plots) and analytical methods (Kolmogorov-Smirnov test). When comparing control and intervention groups, independent groups t-test will be used for comparisons between normally distributed continuous variables, and chi-square test will be used for categorical variables. Comparing the scale scores before and after the application in the intervention group, if the data shows a normal distribution, paired t test will be applied, if it does not show a normal distribution, the Wilcoxon test will be applied. The relationships between variables will be evaluated using Pearson correlation analysis for normally distributed values, and Spearman correlation analysis for non-normally distributed values. Statistical significance level will be accepted as p<0.05

ELIGIBILITY:
Inclusion Criteria:

Being a second year student in the nursing department Not having received training on WEB tools Taking the basic principles and practices course in nursing

Exclusion Criteria:

* Not being a second-year student in the nursing department Having training on WEB tools Not taking the basic principles and practices course in nursing

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Web Pedagogical Content Knowledge Scale: | 6 months
  Web Pedagogical Content Knowledge Scale , consisting of five dimensions and 30 items. Sub-dimensions of the scale created in 5-point Likert type; It has been named as "general web", "communicative web", "pedagogical web", "web pedagogical content", "attitude towards web-based teaching". Cronbach's alpha internal consistency coefficient for the Turkish form was found to be .94. The reliability of the scale was examined with the Cronbach alpha internal consistency coefficient and this value was found to be 0.96 for the entire scale and 0.94, 0.96, 0.94, 0.95 and 0.92 for the factors, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Yasemin Erden, Study Director — Erzurum Technical University Faculty of Health Science
Locations (1):
- Erzurum Technical University, Erzurum, Turkey (Türkiye)